CLINICAL TRIAL: NCT01180348
Title: Randomized Study of Clinical Non-inferiority of Medicine Botulift (Laboratório Químico Farmacêutico Bergamo Ltd.) Compared to Botox ® (Allergan Inc.) in the Improvement of Wrinkles in the Facial Region.
Brief Title: Efficacy and Safety of a New Botulinum Toxin Type A for Treatment of Facial Expression Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Laboratório Químico Farmacêutico Bergamo Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOXBER0610
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Wrinkles
Keywords: Wrinkles, glabellar, facial.
MeSH Terms: conditions — Facies | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulift (Experimental): Application of 90 U of Botulift divided in 3 applications on each side of the face in fifteen predetermined sites in three regions of the face (front, glabellar, periocular).
  Interventions: Drug: Botulift
- Botox (Active Comparator): Application of 90 U of Botox divided in 3 applications on each side of the face in fifteen predetermined sites in three regions of the face (front, glabellar, periocular).
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botulift — Application of 90 U of Botulift divided in 3 applications on each side of the face in fifteen predetermined sites in three regions of the face (front, glabellar, periocular).
  Other Names: Botulinum Toxin Type A
  Arms: Botulift
Drug: Botox — Application of 90 U of Botox divided in 3 applications on each side of the face in fifteen predetermined sites in three regions of the face (front, glabellar, periocular).
  Other Names: Botulinum Toxin Type A
  Arms: Botox

SUMMARY:
The dermatological treatment for reducing facial wrinkles with injectable drug Botulift (botulinum toxin type A - Laboratório Químico Farmacêutico BergamoLtd.) has a not inferior activity when compared with Botox ® (botulinum toxin - Allergan Inc.) in clinical trials.

DETAILED DESCRIPTION:
The study will evaluate non-inferiority in clinical improvement in the intensity of expression lines over 16 weeks of drug Botulift (Laboratório Químico Farmacêutico Bergamo Ltd.) compared with Botox ® (Allergan Inc.). So that the homogeneity of the group opted to use in female patients with glabellar wrinkles grade 2 (moderate) and 3 (severe) Scale Standard Facial Wrinkles, established by Honecker et al. (2003). The first area of the face perceived in mime is the glabellar complex, located in the space between the eyebrows, wrinkles eventually show (Almeida et al., 2010).

Patients will be evaluated at each visit, the doctor Principal Investigator and digital photos of the glabellar region at maximum contraction and relaxation will be obtained using the apparatus Visia (Canfield Imaging Systems, version 4.0.2) for further analysis by random team dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all study procedures and sign for their own free will the TCLE;
* Adult patients were female between 18 and 65 years, regardless of social condition;
* between skin phototype I and IV;
* With good mental and physical health;
* Patients who have not been treated with botulinum toxin type A;
* Patients who agree to abstain from physical activity for a period of 24 hours, previous and subsequent to the initiation of the study;
* Patients presenting at screening visit, wrinkles in the glabellar region between classes 2 and 3 of Table Wrinkles Pattern Classification, which is diagnosed clinically by the dermatologist.

Exclusion Criteria:

* Patients who are in classes 0 and 1 of the Table Pattern Classification Wrinkle;
* Patients who have disorders or diseases that might interfere with neuromuscular function (myasthenia gravis or Lambert-Eaton syndrome);
* Patients being treated with antibiotics (aminoglycosides) and muscle relaxants;
* Patients with pre-existing conditions such as ptosis or scars in the area to be assessed, as they may endanger the health of the patient and the results of the study;
* Patients who have made treatments fill in the glabellar region (retinoic acid, collagen);
* Patients who have been treated in the dermatological peeling úlitmos three months;
* Patients are using treatments dermacosmetics agents anti age (vitamin C pure retinoids flavanoids acid hyaluronic others) or used past 3 months
* Patients with known hypersensitivity to any component of the study drug;
* Pregnant or lactating women;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
overall improved assessment of hyperkinetic facial lines in a state of relaxation and maximal contraction through the Honeck's scale and photographic images obtained by equipment Visia Digital Compexton Analysis (Canfield Imaging Systems, version 4.0.2) | after 30 days of application
  The non-inferiority of T group compared to the group Co was demonstrated in evaluations in a state of relaxation and maximal contraction in the PP analysis population, because as defined for the study, the lower limits of 95% of the mean of these assessments (-2 , 7% and -5.4%) are contained within the non-inferiority limit set at -10%.

SECONDARY OUTCOMES:
Length of stay of the effect of botulinum toxin A (Test and Comparator) | during the 24-week period
  The action of both treatments decreases over time and there is no significant difference between the two treatments.
Safety of both botulinum toxin A | during the whole period
  The occurrence of adverse events was similar in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Regina M. Doi, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda; Alexandre Frederico, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study data will be maked available after journal's approbation. The manuscript contained all of data it has been submitted.

REFERENCES:
- [Background] Jankovic J, Brin MF. Botulinum toxin: historical perspective and potential new indications. Muscle Nerve Suppl. 1997;6:S129-45. PMID 9826986
- [Background] Nigam PK, Nigam A. Botulinum toxin. Indian J Dermatol. 2010;55(1):8-14. doi: 10.4103/0019-5154.60343. PMID 20418969
- [Background] Yang GH, Jung HH. A new botulinum toxin potentially bioequivalent to onabotulinumtoxinA: are there any differences at all? Dermatol Surg. 2013 Jan;39(1 Pt 2):165-70. doi: 10.1111/dsu.12073. No abstract available. PMID 23301820
- [Background] Zagui RM, Matayoshi S, Moura FC. [Adverse effects associated with facial application of botulinum toxin: a systematic review with meta-analysis]. Arq Bras Oftalmol. 2008 Nov-Dec;71(6):894-901. doi: 10.1590/s0004-27492008000600027. Portuguese. PMID 19169530
- [Background] Sposito MMM. Toxina botulínica do tipo A: mecanismo de ação. Acta Fisiatr. 2009;16(1):25-37.
- [Background] Carruthers JA, Lowe NJ, Menter MA, Gibson J, Nordquist M, Mordaunt J, Walker P, Eadie N; BOTOX Glabellar Lines I Study Group. A multicenter, double-blind, randomized, placebo-controlled study of the efficacy and safety of botulinum toxin type A in the treatment of glabellar lines. J Am Acad Dermatol. 2002 Jun;46(6):840-9. doi: 10.1067/mjd.2002.121356. PMID 12063480
- [Background] Small R. Botulinum toxin injection for facial wrinkles. Am Fam Physician. 2014 Aug 1;90(3):168-75. PMID 25077722
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Hexsel D, Mazzuco R, Dal'Forno T, Kraemer C, Lima MM, Prado DZ. Botulinum toxin for Facial Wrinkles: History and Future. Expert Rev. Dermatol. 2(4), 417 - 426 (2007).
- [Background] Carruthers JD, Lowe NJ, Menter MA, Gibson J, Eadie N; Botox Glabellar Lines II Study Group. Double-blind, placebo-controlled study of the safety and efficacy of botulinum toxin type A for patients with glabellar lines. Plast Reconstr Surg. 2003 Sep 15;112(4):1089-98. doi: 10.1097/01.PRS.0000076504.79727.62. PMID 12973229
- [Background] De Boulle K, Fagien S, Sommer B, Glogau R. Treating glabellar lines with botulinum toxin type A-hemagglutinin complex: a review of the science, the clinical data, and patient satisfaction. Clin Interv Aging. 2010 Apr 26;5:101-18. doi: 10.2147/cia.s9338. PMID 20458348
- [Background] Carruthers A, Carruthers J, Cohen J. A prospective, double-blind, randomized, parallel- group, dose-ranging study of botulinum toxin type a in female subjects with horizontal forehead rhytides. Dermatol Surg. 2003 May;29(5):461-7. doi: 10.1046/j.1524-4725.2003.29114.x. PMID 12752512
- [Background] Honeck P, Weiss C, Sterry W, Rzany B; Gladys study group. Reproducibility of a four-point clinical severity score for glabellar frown lines. Br J Dermatol. 2003 Aug;149(2):306-10. doi: 10.1046/j.1365-2133.2003.05436.x. PMID 12932236
- [Background] Dolly, JO. Therapeutic and Research Exploitation of Botulinum Neurotoxins. Eur J Neurol. 1997;4:S5-10.
- [Background] Yoon JS, Kim JC, Lee SY. Double-blind, randomized, comparative study of Meditoxin versus Botox in the treatment of essential blepharospasm. Korean J Ophthalmol. 2009 Sep;23(3):137-41. doi: 10.3341/kjo.2009.23.3.137. Epub 2009 Sep 8. PMID 19794937
- [Background] Kim K, Shin HI, Kwon BS, Kim SJ, Jung IY, Bang MS. Neuronox versus BOTOX for spastic equinus gait in children with cerebral palsy: a randomized, double-blinded, controlled multicentre clinical trial. Dev Med Child Neurol. 2011 Mar;53(3):239-44. doi: 10.1111/j.1469-8749.2010.03830.x. Epub 2010 Nov 18. PMID 21087238
- [Background] Wollmer MA, de Boer C, Kalak N, Beck J, Gotz T, Schmidt T, Hodzic M, Bayer U, Kollmann T, Kollewe K, Sonmez D, Duntsch K, Haug MD, Schedlowski M, Hatzinger M, Dressler D, Brand S, Holsboer-Trachsler E, Kruger TH. Facing depression with botulinum toxin: a randomized controlled trial. J Psychiatr Res. 2012 May;46(5):574-81. doi: 10.1016/j.jpsychires.2012.01.027. Epub 2012 Feb 24. PMID 22364892
- [Background] Ascher B, Rzany BJ, Grover R. Efficacy and safety of botulinum toxin type A in the treatment of lateral crow's feet: double-blind, placebo-controlled, dose-ranging study. Dermatol Surg. 2009 Oct;35(10):1478-86. doi: 10.1111/j.1524-4725.2009.01261.x. Epub 2009 Jul 20. PMID 19686365
- [Background] Beer KR. Comparative evaluation of the safety and efficacy of botulinum toxin type A and topical creams for treating moderate-to-severe glabellar rhytids. Dermatol Surg. 2006 Feb;32(2):184-97. doi: 10.1111/j.1524-4725.2006.32036.x. PMID 16442037
- [Background] Jones D, Carruthers J, Narins RS, Coleman WP 3rd, Harrington L, Brandt FS, Cohen JL. Efficacy of incobotulinumtoxinA for treatment of glabellar frown lines: a post hoc pooled analysis of 2 randomized, placebo-controlled, phase 3 trials. Dermatol Surg. 2014 Jul;40(7):776-85. doi: 10.1111/dsu.0000000000000001. PMID 25111351
- [Background] Won CH, Lee HM, Lee WS, Kang H, Kim BJ, Kim WS, Lee JH, Lee DH, Huh CH. Efficacy and safety of a novel botulinum toxin type A product for the treatment of moderate to severe glabellar lines: a randomized, double-blind, active-controlled multicenter study. Dermatol Surg. 2013 Jan;39(1 Pt 2):171-8. doi: 10.1111/dsu.12072. PMID 23301821
- [Background] RDC 55 - Agência Nacional de Vigilância Sanitária. Registro de Produtos Biológicos | Bases Legais e Guias - Coletânea -459p.: il.; graf.; tab. ISBN.
- [Background] Ferreira LM, Filho ST, Costa RO, Godoy A, Steiner D, Fleissig L, et al. Eficácia e tolerabilidade de uma nova toxina botulínica tipo A para tratamento estético de rugas faciais dinâmicas: estudo multicêntrico prospectivo de fase III. Surgical & Cosmetic Dermatology 2009;1(2): 58-63.
- [Background] Filho ST, Bagatin E, Monteiro EO, Pinheiro MVB, Hassun KM. Eficácia e segurança da neurotoxina botulínica tipo A* no tratamento de linhas de expressão glabelares. RBM rev. bras. med;65(n.esp):28-33, out. 2008.
- [Background] Rappl T, Parvizi D, Friedl H, Wiedner M, May S, Kranzelbinder B, Wurzer P, Hellbom B. Onset and duration of effect of incobotulinumtoxinA, onabotulinumtoxinA, and abobotulinumtoxinA in the treatment of glabellar frown lines: a randomized, double-blind study. Clin Cosmet Investig Dermatol. 2013 Sep 24;6:211-9. doi: 10.2147/CCID.S41537. eCollection 2013. PMID 24098087
- [Background] Gracies JM, Simpson DM. Botulinum toxin therapy. Neurologist 6:98,2000.